CLINICAL TRIAL: NCT06041711
Title: COMPARISON OF THE EFFECTS OF GENERAL AND REGIONAL ANESTHESIA ON SLEEP QUALITY IN PATIENTS PLANNING TOTAL HIP ARTROPLASTY
Brief Title: GENERAL vs. REGIONAL ANESTHESIA ON SLEEP QUALITY FOR HIP ARTROPLASTY PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Elifgül Ulutaş, Research assistant, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-KAEK-26
Record Dates: First submitted 2023-08-30; First posted 2023-09-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-09

CONDITIONS: Sleep Disturbance; Postoperative Complications; Regional Anesthesia Morbidity
MeSH Terms: conditions — Parasomnias; Postoperative Complications | interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator completing the questionnaires will not be aware of patient group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia group (Active Comparator): Patients allocated to the general anesthesia group will be subjected to general anesthesia with induction with propofol and will sevoflurane (inhalational agent) used for maintenance. End of the procedure all patients will be extubated and awakened in the operating room. İntravenous morphine patient-controlled analgesia will be used in the postoperative period.
  Interventions: Procedure: General anesthesia with propofol induction and sevoflurane maintenance
- Regional anesthesia group (Active Comparator): Patients allocated to the regional anesthesia group will be subjected to combined spinal-epidural anesthesia with heavy bupivacaine or spinal anesthesia with PENG(pericapsular nerve group) block with bupivacaine. If lumbar combined spinal epidural anesthesia is applied epidural patient-controlled analgesia will be used in the postoperative period. If spinal anesthesia and PENG block is applied, intravenous morphine patient-controlled analgesia will be used in the postoperative period.
  Interventions: Procedure: Regional anesthesia with neuroaxial blockage

INTERVENTIONS:
Procedure: General anesthesia with propofol induction and sevoflurane maintenance — Surgical procedure is performed under general anesthesia with propofol induction and mainteined with sevoflurane inhalation.
  Arms: General anesthesia group
Procedure: Regional anesthesia with neuroaxial blockage — Surgical procedure is performed under regional anesthesia. Patients are sedated with 2 mg intravenous midazolam. Combined spinal epidural anesthesia or spinal anesthesia with PENG block is used for anesthesia and analgesia.
  Arms: Regional anesthesia group

SUMMARY:
Sleep disorders can impair cognitive function, decision-making ability, exercise capacity, and immune system.Sleep disorders, which may occur in the perioperative period as short-term or long-term, affect many patients. Patients have to face with perioperative sleep disorders, and this situation can continue for a long time after surgery.

Anesthetic agents may cause sleep disturbances in the postoperative period. Anesthetics can disrupt the normal sleep-wake cycle and thus cause sleep insufficiency and poor sleep quality. The relationship between general anesthesia and postoperative sleep disorders is still unclear. It is advantageous to identify patients with pre-existing sleep disorders, since the risk of postoperative sleep disturbance is high.

The investigators hypothesis that regional anesthesia does not disrupt the circadian rhythm compared to general anesthesia, is more successful in pain control, and thus provides a better sleep quality for patients.

DETAILED DESCRIPTION:
Sleep is one of the basic physiological needs of man and is necessary for the normal functioning of the body. Sleep disorders can impair cognitive function, decision-making ability, exercise capacity, and immune system. Sleep disorders, which may occur in the perioperative period as short-term or long-term, affect many patients. Studies have shown that approximately 8.8-79.1% of patients experience perioperative sleep disorders, and this situation can continue for a long time after surgery.

According to animal and human studies, anesthetic agents may cause sleep disturbances in the postoperative period. Anesthetics can disrupt the normal sleep-wake cycle and thus cause sleep insufficiency and poor sleep quality. Since postoperative pain and emotional changes will also cause sleep disturbances, the view that general anesthesia impairs postoperative sleep quality has not yet been proven.

Pain is the most important risk factor for sleep disturbance in the perioperative period. There is a very serious interaction between pain and sleep. Pain can exacerbate sleep disorders. At the same time, sleep disorders can make the pain worse. Perioperative pain accompanies physical discomfort and is very common, especially in osteoarthritis patients. The goals of total hip arthroplasty (TKA) include relief of these pains and improvement of physical function.

Different types of surgery have varying effects on sleep quality. Patients report that they experience more sleep disruption due to pain after orthopedic surgery. Depending on the greater trauma caused by major surgery, the sleep quality of the patients may be worse.

The elderly and female gender are more likely to experience sleep disorders. Environmental factors and healthcare practices in the hospital may contribute to sleep disorders. Postoperative environment change, inadequate beds, noise and lights in the ward, medical staff, night treatment and nursing controls, machine noises, postoperative diets and warnings from the urinary catheter are additional factors that affect patients' sleep.

Evaluation of sleep disorders is mainly based on clinical symptoms (difficulty falling asleep, early awakening, night terrors, nightmares or abnormal behavior during the sleep period) and auxiliary objective scales. Subjective sleep quality assessment mainly scales: Pittsburgh Sleep Quality Index questionnaire (PSQI), Pittsburgh Insomnia Rating Scale (PIRS), Insomnia Severity Index (ISI), Athens Insomnia Scale, Epworth Sleepiness Scale (ESS), General Sleep Disturbance Scale (GSDS). It is in the form. The most commonly used assessment in clinical studies is the PSQI. PSQI has high reliability and validity, but evaluates over a one-month period. The PIRS_20 scale, which is a self-assessment survey, is a scale created by the Department of Psychiatry at the University of Pittsburgh and evaluates the participants' sleep quality in the last week. It generally consists of a questionnaire with a total of twenty items, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disorders. Scoring ranges from 0 to 60. A score of 20 and above indicates poor sleep quality, while as the score increases, sleep quality deteriorates. As another assessment of sleep quality, the ISI is a self-rating scale that measures insomnia symptoms and consequences. Substances include difficulties in initiating sleep and maintaining sleep; It is designed to assess satisfaction with current sleep patterns, disruption in daily life, cognitive impairments, and the degree of anxiety or worry caused by sleep disturbance. The severity of insomnia is also determined by the total score of these items. Additionally, ESS is used to evaluate the tendency to sleep during the day.

Sleep disorders can negatively impact patient recovery, contributing to higher rates of postoperative complications such as neurological and cardiovascular morbidity and delayed postoperative recovery. They are also risk factors for cardiovascular and cerebrovascular diseases such as myocardial infarction, as well as dementia, obesity, diabetes, hypertension, depression, pain and even death. It is also considered an important risk factor for the development of delirium. Despite posing a significant threat to public health, sleep disorders remain poorly understood, underdiagnosed, and poorly managed, especially in perioperative patients. The potential negative consequences of sleep disorders indicate that more attention should be paid to this issue.

Risk factors that increase sleep problems include postoperative pain, depression, anxiety, and physical disabilities. Sleep problems experienced the night before surgery may affect postoperative pain due to various other factors. has an even more significant effect. Sleep quality assessment is not a part of the pre-anaesthesia routine evaluation of patients and adequate attention is not paid to perioperative management.

The type of anesthesia is also one of the factors on sleep quality. It is known that the anesthesia process (general anesthesia (GA) or regional anesthesia (RA)) affects melatonin rhythm. General anesthetics act centrally on the sleep center, causing sedation, hypnosis, and unconsciousness similar to a dreamless sleep. General anesthesia disrupts the sleep/wake cycle, other circadian rhythms such as body temperature regulation and melatonin secretion.

Regional anesthesia is thought to be more advantageous than general anesthesia in eliminating postoperative sleep disorders.

In this study, changes in sleep patterns and simultaneous changes in sleep patterns caused by regional and general anesthesia in patients who underwent total hip arthroplasty by using PID-20 (Pittsburg Insomnia Rating Scale_20), VAS (Visual Analogue Scale), Wong Baker Pain Scale, Momentary (State) Anxiety Scale scales. We aimed to evaluate anxiety and pain levels.

Despite the importance of sleep quality assessment, it is not a part of the routine pre-anesthesia evaluation of patients and does not receive enough attention. Preoperative sleep assessment can provide information that may allow early intervention by anesthetists. There are no guidelines and sufficient number of studies for clinical use.

Postoperative sleep disorders have serious effects on cognition, pain perception, altered circadian rhythm, psychomotor function, cardiovascular outcomes, metabolic function, catabolic responses, and inflammation. The relationship between general anesthesia and postoperative sleep disorders is still unclear. It is advantageous to identify patients with pre-existing sleep disorders, since the risk of postoperative sleep disturbance is high. The investigators hypothesis that regional anesthesia does not disrupt the circadian rhythm compared to general anesthesia, is more successful in pain control, and thus provides a better sleep quality for patients.

Protocol:

A total of 60 patients whom undergo total hip arthroplasty by Bursa Uludağ University Faculty of Medicine, Department of Orthopedics and Traumatology are included in this study.

Inclusion criteria: 18 years of age and older, score between I and III according to the American Society of Anesthesiologists (ASA) classification.

Exclusion criteria : Patients who underwent THA with urgent indication, patients under 18, ASA score 4 and above, patients who do not accept informed consent, those who refuse to participate in the study Patients are evaluated for sleep quality with the PID-20 (Pitssburg Insomnia Rating Scale) at least 1 month before the surgery date, and re-evaluated the night before and 1 week after the surgery. During this process, patients evaluated simultaneously with the VAS (Visual Analogue Scale), Wong Baker Pain Scale and Immediate (State) Anxiety Scale. The relationship between pain and anxiety and sleep quality are evaluated.

Patients are monitored in terms of possible complications, mortality and morbidity in the postoperative 3 months.

All evaluations are performed in the hospital where the patient is hospitalized and by the same anesthesiologist for a standard evaluation.

Demographic information (name-surname, protocol number, age, co-morbidity, medications used, habits, ASA score) of the patients are recorded. After the necessary information is given to the patients, their written and verbal consent is obtained.

Routine monitoring (electrocardiography, invasive/noninvasive blood pressure measurement, arterial blood gas monitoring, peripheral oxygen saturation, end-tidal carbon dioxide measurement with capnograph) are applied to the patients in the operating room in accordance with the standard protocol for elective total hip arthroplasty surgery, the anesthetic and analgesic drugs administered are recorded and hemodynamic changes in the intraoperative period (dysrhythmia, hypotension, hypertension), intraoperative complications (transfusion need, allergic reactions, etc.) are recorded. If lumbar combined spinal epidural anesthesia is applied for the regional anesthesia group, epidural patient-controlled analgesia is used in the postoperative period; If spinal anesthesia is applied, an additional PENG (pericapsular nerve group block) block is performed with the help of ultrasound and intravenous morphine patient-controlled analgesia used in the postoperative period. The general anesthesia group is extubated and awakened in the operating room, and intravenous morphine patient-controlled analgesia is used in the postoperative period.

In the postoperative period, intensive care unit stay, duration of hospital stay, early complications (pain, mobilization problems, hypertension, anxiety disorder, dysrhythmia, acute coronary syndrome, sepsis, pneumonia, infections, etc.) is followed up in the postoperative 3 months period.

ELIGIBILITY:
Inclusion Criteria:

* Planning of total hip arthroplasty (primary/redo)
* Elective procedure planning
* 18 years and older patients
* ASA score between I-III
* Approved and signed the informed consent form

Exclusion Criteria:

* Patients who underwent THA with urgent indication
* Patients under 18 years of age
* Patients with ASA score 4 and above
* Patients who do not accept informed consent
* Those who refuse to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality (evaluated by PIRS-20 (Pitssburg Insomnia Rating Scale)) | preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Sleep quality evaluated by PIRS-20 (Pitssburg Insomnia Rating Scale) , a scale provides ranging from 0 to 60 , with a high score indicating a poor quality of sleeping.

SECONDARY OUTCOMES:
Subjective anxiety level | Preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Anxiety level evaluated by STAI (The State Trait Anxiety Inventory), a scale provides ranging from 20 to 80, with a high score indicating high levels of anxiety.
Subjective pain level | Preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Pain level evaluated by VAS (Visuel analog scale) , a scale provides ranging from 0 to 10, with a high score indicating high levels of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ University Faculty of Medicine, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided